CLINICAL TRIAL: NCT04243499
Title: A First-in-human, Two-part Clinical Study to Assess the Safety, Tolerability and Activity of IV Doses of ICT01 as Monotherapy and in Combination With a Checkpoint Inhibitor, in Patients With Advanced-stage, Relapsed/Refractory Cancer
Brief Title: First-in-Human Study of ICT01 in Patients With Advanced Cancer
Acronym: EVICTION
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: ImCheck Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ICT01-101
Record Dates: First submitted 2020-01-24; First posted 2020-01-28 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Solid Tumor, Adult; Hematopoietic/Lymphoid Cancer
Keywords: gamma delta T cells; butyrophilin; pembrolizumab
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Intervention Model Description: Patients will be assigned to a dose level of ICT01 at the time of their enrollment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- IV ICT01 Monotherapy (Experimental): Up to six ICT01 dose levels administered as IV monotherapy every 3 weeks will be tested in Part 1 Dose Escalation and up to 2 dose levels in Part 2 Cohort Expansion
  Interventions: Biological: IV ICT01
- IV ICT01 + IV Pembrolizumab (Experimental): A range of IV ICT01 doses administered every 3 weeks will be tested in combination with 200 mg pembrolizumab in Part 1 Dose Escalation and up to 2 dose levels of ICT01 plus 200 mg pembrolizumab in Part 2 Cohort Expansion
  Interventions: Biological: IV ICT01

INTERVENTIONS:
Biological: IV ICT01 — humanized anti-Butyrophilin 3A (BTN3A) monoclonal antibody

SUMMARY:
Part 1 will be a dose escalation study of IV ICT01 (a monoclonal antibody targeting BTN3A) as monotherapy in patients with advanced solid or hematologic tumors, followed by a cohort examining the combination of ICT01 plus pembrolizumab (Keytruda). Part 2 will be a cohort expansion into 2 solid tumor indications and one hematologic malignancy for ICT01 monotherapy, and 3 solid tumor indications for the combination of ICT01 plus pembrolizumab.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily signed informed consent form.
2. Relapsed/refractory patients with histologically or cytologically confirmed diagnosis of advanced-stage or recurrent cancer, including:

   Group A: bladder, breast, colon, gastric, melanoma, ovarian, prostate and PDAC Group B: hematologic malignancies including acute myeloid leukemia, acute lymphocytic leukemia, Diffuse large B cell lymphoma and follicular lymphoma Group C: melanoma, cervical, bladder, gastric, head and neck SCC, and lymphoma (according to the approved package labeling of the ICI) Part 2, Group D: Ovarian cancer (2L/3L) with baseline g9d2 T cells > 20K Part 2, Group E: metastatic castrate resistant prostate cancer (2L/3L) with baseline g9d2 T cells > 20K Part 2, Group F: newly diagnosed AML starting venetoclax/azacitidine Part 2, Group G: checkpoint-refractory metastatic melanoma with g9d2 T cells >5K Part 2, Group H: chemotx-refractory or Pt-ineligible urotherlial cancer (bladder) with g9d2 T cells >5K Part 2, Group I: checkpoint-refractory, metastatic HNSCC with g9d2 T cells >5K
3. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1
4. Life expectancy > 3 months as assessed by the Investigator
5. At least 1 measurable lesion per Response Evaluation Criteria in Solid Tumors (RECIST)/ Response Evaluation Criteria in Lymphoma (RECIL) or >5% marrow blasts

Exclusion Criteria:

1. Any malignancy of Vγ9Vδ2 T cell origin
2. Any anti-tumor-directed drug therapy within 28 days or 5 times the elimination half-life (whichever is shorter) before study treatment (does not apply to patients receiving ICI for the combination arm)
3. Treatment with investigational drug(s) within 28 days before study treatment
4. Systemic steroids at a daily dose of > 10 mg of prednisone, > 2 mg of dexamethasone or equivalent, for the last 28 days and need for ongoing treatment.
5. Patients with rapidly progressing disease defined as advanced/metastatic, symptomatic, visceral spread, with a risk of life-threatening complications in the short term (e.g., during Screening Period/ treatment washout) that includes patients with massive uncontrolled effusions pleural, pericardial, peritoneal, pulmonary lymphangitis, and over 50% liver involvement
6. Ongoing immune-related adverse events (irAEs) and/or AEs ≥grade 2 not resolved from previous therapies except vitiligo, stable neuropathy up to grade 2, hair loss, and stable endocrinopathies with replacement hormone therapy.
7. Within 4 weeks of major surgery
8. Documented history of active autoimmune disorders requiring systemic immunosuppressive therapy within the last 12 months
9. Primary or secondary immune deficiency
10. Active and uncontrolled infections requiring intravenous antibiotic or antiviral treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 292 (Actual)
Dates: Start 2020-03-05 (Actual); Primary Completion 2025-10-15 (Actual); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Adverse Events (Parts 1 & 2) | 12 months
  Incidence of treatment-emergent adverse events
Disease Control Rate using RECIST for solid tumor patients (Part 2) | 12 months
  RECIST is measured every 8 weeks during treatment
Disease Control Rate using RECIL for lymphoma patients (Part 2) | 12 months
  RECIL is measured every 8 weeks during treatment

SECONDARY OUTCOMES:
Change from Baseline in the Number of Circulating Gamma Delta T Cells | 28 days
  Flow cytometric counting of circulating gamma delta T cells
Change from Baseline in the Activation State of Circulating Gamma Delta T Cells | 28 days
  Flow cytometric measurement of CD69 and Ki67 expression on gamma delta T cells
Cmax following the first dose of ICT01 | 1 day
  PK parameter from serum ICT01 levels
AUC following the first dose of ICT01 | 21 days
  PK parameter from serum ICT01 levels
Clearance at steady-state of ICT01 | 6 months
  PK parameter from serum ICT01 levels
Half-life of ICT01 | 6 months
  PK parameter from serum ICT01 levels
Objective Response Rate using RECIST for solid tumor patients (Part 2) | 12 months
  RECIST is measured every 8 weeks during treatment

CONTACTS AND LOCATIONS:
Overall Officials: Katrien Lemmens, MD, PhD, Study Director — ImCheck Therapeutics
Locations (29):
- United States (8):
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Yale Cancer Center, New Haven, Connecticut
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Montefiore Medical Center, The Bronx, New York
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - US Oncology Research, Irving, Texas
  - University of Washington, Seattle, Washington
- Institut Jules Bordet, Brussels, Belgium
- France (12):
  - Institut Bergonie, Bordeaux
  - Haut Leveque, Bordeaux
  - Centre Hospitalier Lyon Sud, Lyon
  - Centre Lyon Berard, Lyon
  - CHU Lyon, Lyon
  - Institut Paoli-Calmettes, Marseille
  - CHU Nantes, Nantes
  - Centre Antoine Lacassagne, Nice
  - Pitie-Salpetriere, Paris
  - Institut Curie, Paris
  - Gustave Roussy, Paris
  - CHU Poitiers, Poitiers
- Germany (2):
  - University Carl Gustav Carus Clinical Trial Unit, Dresden
  - universitatklinikum Wurburg, Würzburg
- Spain (4):
  - START Barcelone HM Nou Delfos, Barcelona
  - Vall d'Hebron Instiute of Oncology, Barcelona
  - START Madrid-FJD, Hospital Fundación Jiménez Díaz, Madrid
  - Hospital Universitario HM Sanchinarro, Madrid
- United Kingdom (2):
  - NHS Greater Glasgow and Clyde, Beatson West of Scotland Cancer Centre, Glasgow
  - Institute of Cancer Research, London

IPD SHARING:
Plan to Share IPD: No